CLINICAL TRIAL: NCT00751803
Title: A Randomised, Double-blind, Placebo- and Active Comparator-controlled, Five Parallel Groups Study to Investigate the Efficacy and Safety of BI 44370 TA (50 mg, 200 mg, and 400 mg) Administered Orally Once During an Acute Migraine Attack of Moderate or Severe Intensity
Brief Title: BI 44370 TA in Acute Migraine Attack
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 1246.4; EudraCT No : 2008-000079-31
Record Dates: First submitted 2008-08-25; First posted 2008-09-12 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-11

CONDITIONS: Migraine Disorders
MeSH Terms: conditions — Migraine Disorders | interventions — eletriptan

ARMS (5):
- BI 44370 TA Low Dose (Experimental)
  Interventions: Drug: BI 44370 TA Low Dose; Drug: Placebo
- BI 44370 TA Medium Dose (Experimental)
  Interventions: Drug: Placebo; Drug: BI 44370 TA Medium Dose
- BI 44370 TA High Dose (Experimental)
  Interventions: Drug: Placebo; Drug: BI 44370 TA Medium Dose
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Eletriptan (Active Comparator)
  Interventions: Drug: Eletriptan; Drug: Placebo

INTERVENTIONS:
Drug: BI 44370 TA Low Dose
  Arms: BI 44370 TA Low Dose
Drug: Eletriptan
  Arms: Eletriptan
Drug: Placebo
Drug: BI 44370 TA Medium Dose
  Arms: BI 44370 TA High Dose; BI 44370 TA Medium Dose

SUMMARY:
The objective of this trial is to assess the safety, tolerability, and efficacy of three doses of BI 44370 TA in the treatment of patients with an acute migraine attack and headache pain of moderate or severe intensity, compared to placebo and an active comparator.

ELIGIBILITY:
Inclusion Criteria:

* Adult migraine patients with or without aura, diagnosed according to the ICH.
* Established migraine diagnosis greater than or equal to 1 year.
* Age at first migraine onset latest at 50 years of age.
* Medical history of migraine with headache of moderate to severe intensity and migraine frequency of 2-8 times/ month.
* Patient has provided written informed consent in accordance with ICH-GCP and local legislation.

Exclusion Criteria:

* History of hemiplegic, ophthalmoplegic or basilar migraine, or cluster headache.
* History of treatment-resistant migraine attacks.
* Other pain syndromes possibly interfering with study assessment or use of any pain medication > 10 days / month.
* Use of migraine and other restricted medication, or other restrictions as per protocol.
* Pregnancy or breast-feeding. Female of childbearing potential who do not use contraception.
* Clinically significant cardiovascular, peripheral vascular, hepatic, respiratory, haematological, gastrointestinal, renal, metabolic, immunological, hormonal, neurological and psychiatric disorders.
* Patients in whom unrecognised coronary artery disease is likely, or who are at risk of coronary artery disease indicated by the presence of risk factors.
* Persistent liver enzyme elevation such as ALT, AST or AP > 2x ULN.
* Known history of HIV, or history of cancer within the last 5 years.
* DSM-IV-defined-history of substance abuse or dependence within the past 6 months, excluding nicotine and caffeine, but including alcohol or benzodiazepines.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Actual)
Dates: Start 2008-08; Primary Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is a pain free response, defined as reduction of severe or moderate headache to no headache, 2 hours after dosing. | 2 hours

SECONDARY OUTCOMES:
Pain-free response 0.5, 1, 1.5, 24 and 48 hours after dosing | up to 48 h
Pain relief, defined as reduction of severe or moderate headache to mild or no headache, 0.5, 1, 1.5, 2, 24 and 48 hours after dosing | up to 48 h
Sustained pain-free response, defined as reduction of severe or moderate headache to no headache 2 hours after dosing and remaining pain-free up to 24 and 48 hours after dosing | up to 48 h
Sustained pain relief response, defined as reduction of severe or moderate headache to mild or no headache 2 hours after dosing and no worsening up to 24 and 48 hours after dosing | up to 48 h
Intensity of headache at the time of intake of study medication, and 0.5, 1, 1.5, 2, 24 and 48 hours after dosing | up to 48 h
Relief of associated migraine symptoms (nausea, vomiting, photophobia, phonophobia) 0.5, 1, 1.5, 2, 24 and 48 hours after dosing | up to 48 h
Time to meaningful relief, defined by the patient as occurring when relief of pain and associated symptoms becomes meaningful, up to 2 h after dosing | up to 2 h
Global evaluation of medication by the patient evaluated 48 h after study drug intake | up to 48 h
Functional disability assessed by the patient measured at the time of intake of study medication, and 0.5, 1, 1.5, 2, 24 and 48 hours post dosing | up to 48 h
Time to and use of rescue medication within 24 and 48 hours | up to 48 h
Recurrence / relapse of headache during time-intervals of 2-24 and 2-48 hours post dosing | up to 48 h
Incidences of adverse events | up to 7 days
Changes from baseline in safety laboratory parameters | up to 7 days
Changes from baseline in vital sign parameters | up to 7 days
Withdrawals due to adverse events | up to 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (52):
- Belgium (8):
  - 1246.4.32004 Boehringer Ingelheim Investigational Site, Antwerp
  - 1246.4.32005 Boehringer Ingelheim Investigational Site, Brussels
  - 1246.4.32006 Boehringer Ingelheim Investigational Site, Charleroi
  - 1246.4.32001 Boehringer Ingelheim Investigational Site, Ghent
  - 1246.4.32002 Boehringer Ingelheim Investigational Site, Hasselt
  - 1246.4.32009 Boehringer Ingelheim Investigational Site, Leuven
  - 1246.4.32007 Boehringer Ingelheim Investigational Site, Liège
  - 1246.4.32008 Boehringer Ingelheim Investigational Site, Montegnée
- 1246.4.34004 Boehringer Ingelheim Investigational Site, Oviedo, El Salvador
- France (10):
  - 1246.4.3307A Boehringer Ingelheim Investigational Site, Clermont-Ferrand
  - 1246.4.3307B Boehringer Ingelheim Investigational Site, Clermont-Ferrand
  - 1246.4.3303A Boehringer Ingelheim Investigational Site, Lille
  - 1246.4.3301A Boehringer Ingelheim Investigational Site, Nice
  - 1246.4.3301B Boehringer Ingelheim Investigational Site, Nice
  - 1246.4.3305B Boehringer Ingelheim Investigational Site, Paris
  - 1246.4.3304A Boehringer Ingelheim Investigational Site, Rouen
  - 1246.4.3304B Boehringer Ingelheim Investigational Site, Rouen
  - 1246.4.3302A Boehringer Ingelheim Investigational Site, Toulouse
  - 1246.4.3302B Boehringer Ingelheim Investigational Site, Toulouse
- Germany (10):
  - 1246.4.49002 Boehringer Ingelheim Investigational Site, Berlin
  - 1246.4.49003 Boehringer Ingelheim Investigational Site, Erkelenz
  - 1246.4.49001 Boehringer Ingelheim Investigational Site, Essen
  - 1246.4.49006 Boehringer Ingelheim Investigational Site, Göttingen
  - 1246.4.49004 Boehringer Ingelheim Investigational Site, Grevenbroich
  - 1246.4.49011 Boehringer Ingelheim Investigational Site, Hüttenberg
  - 1246.4.49007 Boehringer Ingelheim Investigational Site, Koenigstein Im Taurus
  - 1246.4.49008 Boehringer Ingelheim Investigational Site, Munich
  - 1246.4.49009 Boehringer Ingelheim Investigational Site, Munich
  - 1246.4.49010 Boehringer Ingelheim Investigational Site, Münster
- Italy (6):
  - 1246.4.39005 Boehringer Ingelheim Investigational Site, Bologna
  - 1246.4.39006 Boehringer Ingelheim Investigational Site, Catania
  - 1246.4.39001 Boehringer Ingelheim Investigational Site, Milan
  - 1246.4.39004 Boehringer Ingelheim Investigational Site, Milan
  - 1246.4.39003 Boehringer Ingelheim Investigational Site, Roma
  - 1246.4.39002 Boehringer Ingelheim Investigational Site, Torino
- Netherlands (6):
  - 1246.4.31001 Boehringer Ingelheim Investigational Site, 's-Hertogenbosch
  - 1246.4.31004 Boehringer Ingelheim Investigational Site, Amsterdam
  - 1246.4.31003 Boehringer Ingelheim Investigational Site, Blaricum
  - 1246.4.31002 Boehringer Ingelheim Investigational Site, Breda
  - 1246.4.31005 Boehringer Ingelheim Investigational Site, Nijmegen
  - 1246.4.31006 Boehringer Ingelheim Investigational Site, Zwolle
- Spain (3):
  - 1246.4.34002 Boehringer Ingelheim Investigational Site, Barcelona
  - 1246.4.34005 Boehringer Ingelheim Investigational Site, Santiago de Compostela
  - 1246.4.34001 Boehringer Ingelheim Investigational Site, Valencia
- Sweden (4):
  - 1246.4.46001 Boehringer Ingelheim Investigational Site, Gothenburg
  - 1246.4.46004 Boehringer Ingelheim Investigational Site, Linköping
  - 1246.4.46005 Boehringer Ingelheim Investigational Site, Stockholm
  - 1246.4.46002 Boehringer Ingelheim Investigational Site, Vällingby
- United Kingdom (4):
  - 1246.4.44013 Boehringer Ingelheim Investigational Site, Liverpool
  - 1246.4.44001 Boehringer Ingelheim Investigational Site, Oxford
  - 1246.4.44003 Boehringer Ingelheim Investigational Site, Plymouth
  - 1246.4.44007 Boehringer Ingelheim Investigational Site, Whitechapel, London